CLINICAL TRIAL: NCT02159170
Title: Cortical Representation of NGF-induced Hyperalgesia
Brief Title: Cortical Representation of Hyperalgesia Induced by Nerve Growth Factor
Acronym: LOGIN_NGF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof Herta Flor (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Sponsor-Investigator, Prof Herta Flor, Prof. Dr. Herta Flor, Central Institute of Mental Health, Mannheim
Organization: Central Institute of Mental Health, Mannheim (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LOGIN_NGF; 01ED1010D (Other Grant/Funding Number: German Ministry for Education and Research)
Record Dates: First submitted 2014-06-03; First posted 2014-06-09 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Non-inflammatory Neuropathic Pain; Healthy Subjects
Keywords: Use of NGF injection as a model of non-inflammatory neuropathic pain in healthy subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NGF (Experimental): injection of 50 µl NGF, once into the left volar forearm and injection of 50 µl NaCl (sodium chloride) once into the right volar forearm
  Interventions: Biological: NGF injection

INTERVENTIONS:
Biological: NGF injection — single injection of NGF into the volar forearm / single injection of NaCl into the volar forearm

SUMMARY:
Intraepidermal injection of nerve growth factor results in a non-inflammatory hyperalgesia for thermal and mechanical stimuli. This hyperalgesia is similar to the pathological ailments of patients with neuropathic pain. The mechanisms of the cognitive modulation of pain and hyperalgesia are not yet understood in this group of patients. The investigators plan to use NGF injection as a model of non-inflammatory neuropathic pain in healthy subjects to investigate the underlying neuronal mechanisms of this hyperalgesia using functional magnetic resonance imaging and resting state network analysis.

ELIGIBILITY:
Inclusion Criteria:

* no acute or chronic disease
* no acute or chronic pain
* age: 18-60 years
* male
* no medication use

Exclusion Criteria:

* metallic parts in the body
* claustrophobia
* drug or substance abuse

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in activation of the pain processing and resting state networks | baseline to one week
  Activation of the resting state network (using functional magnetic resonance imaging (fMRI) and a standard echo planar imaging (EPI) sequence) as well as acitvation of the pain processing network (using fMRI and a standard EPI sequence) in response to painful stimulation, will be measured before and after injection of NGF into the volar forearm of the participant.
  Particants are measured 0-4 days before injection (baseline) and then again 4-7 days after injection (to measure changes due to NGF injection).

SECONDARY OUTCOMES:
Changes in pain intensity, unpleasentness and suffering ratings | baseline to one week
  Pain will be applied by using impact stimulation to the side where NGF was injected as well as a control side. Pain and tolerance thresholds as well as 3 ratings of intensity/unpleasantness and suffering will be obtained immediately after stimulation.
  This will take place before NGF injection (baseline, 0-4 days) and after NGF injection (4-7 days).
  Ratings will be conducted on visual analog scale from 0 (no pain/unpleasantess/suffering) to 100 (worst pain/unpleasantness/suffering imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Herta Flor, PhD, Principal Investigator — Medical Faculty Mannheim, Heidelberg University
Locations (1):
- Central Institute of Mental Health, Mannheim, Germany